CLINICAL TRIAL: NCT03080974
Title: Immunotherapy and Irreversible Electroporation in the Treatment of Advanced Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Robert C. Martin, Principal Investigator, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16.1190
Record Dates: First submitted 2017-02-14; First posted 2017-03-15 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: irreversible electroporation; Nivolumab
MeSH Terms: interventions — Nivolumab; Electroporation

STUDY DESIGN:
Intervention Model Description: All patients will undergo irreversible electroporation and treatment with Nivolumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): All patients undergoing irreversible electroporation will be treated with nivolumab
  Interventions: Drug: Nivolumab; Procedure: Irreversible Electroporation

INTERVENTIONS:
Drug: Nivolumab — Given post-operatively every two weeks for a total of 4 doses. Dose based on weight.
Procedure: Irreversible Electroporation — Non-thermal ablation of tumor

SUMMARY:
Compare the efficacy and tolerability of irreversible electroporation in combination with Nivolumab in patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Immunotherapy and irreversible electroporation in the treatment of advanced pancreatic adenocarcinoma. This is a Phase II study in which all patients undergoing irreversible electroporation of locally advanced pancreatic adenocarcinoma will be treated with nivolumab post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years if age
* Diagnosed with stage III pancreatic cancer
* Tumor is measurable
* Glomerular Filtration Rate > 60 m/L/min/1.73 m(2)
* Willing and able to comply with the protocol requirements
* Able to comprehend and have signed the informed consent to participate

Exclusion Criteria:

* Participating in another clinical trial for the treatment of cancer at time of screening
* Are pregnant or currently breast feeding
* Have a cardiac pacemaker or Implantable Cardioverter Defibrillator implanted that cannot be deactivated during the procedure
* Have non-removable implants with metal parts within 1 cm of the target lesion
* Had a myocardial infarction within 3 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-08-14 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of Combination Irreversible Electroporation and Nivolumab Treatment | Baseline thru 100 days after receiving last dose
  Adverse events and Serious adverse events will be collected

SECONDARY OUTCOMES:
Progression Free Survival | Every three months for 4 years.
  CT scans will be reviewed
Overall Survival | Every three months for 4 years.
  CT scans will be reviewed

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States